CLINICAL TRIAL: NCT05157841
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of EXPAREL vs. Bupivacaine Hydrochloric Acid (HCl) Administered as a Sciatic (in the Popliteal Fossa) Nerve Block for Postsurgical Analgesia in Subjects Undergoing Bunionectomy
Brief Title: Phase 3, Sciatic Nerve Block With EXPAREL for Subjects Undergoing Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 402-C-334
Record Dates: First submitted 2021-11-15; First posted 2021-12-15 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Bunionectomy; Hallux Valgus
Keywords: EXPAREL; Bupivacaine; Analgesia
MeSH Terms: conditions — Hallux Valgus; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Individuals preparing and administering study drug, or transporting unblinded drug will not be allowed to perform any of the study assessments after randomization (with the possible logistical exception of drawing blood in the operating room (OR) to be processed by blinded staff for the PK assessments) or reveal the assigned study treatment to any other members of the study team at any time. Additionally, efforts will be made to prevent the subject from observing the study drug syringe. Staff members conducting study-specific, postsurgical assessments and the subjects will remain blinded to the assigned treatment throughout the study in part by not being present during the administration of the nerve block. The site PI must be blinded to the study drug and will not be involved in and/or present during study drug administration. No crossover will be permitted between the blinded and unblinded study personnel throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: EXPAREL 266 mg arm (Experimental): subjects randomized to this treatment arm will receive 20 mL (266 mg) EXPAREL mixed with 10 mL saline
  Interventions: Drug: Bupivacaine liposome injectable suspension 266 mg
- Part A: EXPAREL 133 mg arm (Experimental): subjects randomized to this treatment arm will receive 10 mL (133 mg) EXPAREL mixed with 20 mL saline
  Interventions: Drug: Bupivacaine liposome injectable suspension 133 mg
- Part A: Bupivacaine HCl arm (Active Comparator): Subjects randomized to this treatment arm will receive 20 mL (50 mg) 0.25% bupivacaine HCl mixed with 10 mL saline
  Interventions: Drug: Bupivacaine HCl
- Part B: EXPAREL 133 mg arm OR EXPAREL 266 mg arm (Experimental): Subjects randomized to this treatment arm will receive 20 mL (266 mg) EXPAREL mixed with 10 mL saline OR 10 mL (133 mg) EXPAREL mixed with 20 mL saline. Dose will be determined following interim analysis of Part A.
  Interventions: Drug: Bupivacaine liposome injectable suspension 133 mg
- Part B: Bupivacaine HCl arm (Active Comparator): subjects randomized to this treatment arm will receive 20 mL (50 mg) 0.25% bupivacaine HCl mixed with 10 mL saline
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Bupivacaine liposome injectable suspension 266 mg — Sciatic nerve block in the popliteal fossa with EXPAREL 266 mg
  Other Names: EXPAREL
  Arms: Part A: EXPAREL 266 mg arm
Drug: Bupivacaine HCl — Sciatic nerve block in the popliteal fossa with Bupivacaine HCl
  Arms: Part A: Bupivacaine HCl arm; Part B: Bupivacaine HCl arm
Drug: Bupivacaine liposome injectable suspension 133 mg — Sciatic nerve block in the popliteal fossa with EXPAREL 133 mg
  Other Names: EXPAREL
  Arms: Part A: EXPAREL 133 mg arm; Part B: EXPAREL 133 mg arm OR EXPAREL 266 mg arm

SUMMARY:
The study is conducted sequentially in two parts.

Part A: The purpose is to obtain information on pharmacokinetic (PK) profile, pharmacodynamics (PD), efficacy, safety, and to assess the performance of 266 mg EXPAREL vs 133 mg EXPAREL.

Part B: The purpose is to evaluate the efficacy and safety of the preferred dosage of EXPAREL from Part A compared with bupivacaine HCl.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, active controlled study in approximately 180 subjects undergoing bunionectomy. The study will be conducted in two parts (Part A and Part B). Part A will be completed and analyzed before enrollment in Part B is initiated.

Subjects may be screened up to 45 days prior to the day of surgery but eligibility must be re-confirmed on the day of surgery prior to randomization.

The following screening procedures will be performed after the informed consent form (ICF) is signed (if not standard of care): assess eligibility, record medical/surgical history, record prior and concomitant medications, record demographics and baseline characteristics, record subject height and weight for body mass index (BMI) calculation, assess chronic opioid use in the past 30 days, conduct urine pregnancy test for women of childbearing potential, perform 12-lead EKG, record serious adverse events (SAEs) starting when the ICF is signed, and record medications for treatment of SAEs.

On Day 1, prior to sciatic nerve block, study staff will review Pain Rating Guide with the subject and record their responses to:

* Numeric rating scale (NRS) score on the worst pain of their operative foot in the last 30 days.
* NRS score on the average pain of their operative foot in the last 30 days.

Part A will enroll approximately 60 subjects undergoing bunionectomy into 1 of 3 arms. They will be randomized 1:1:1 to either EXPAREL 266 mg, EXPAREL 133 mg, or 0.25% bupivacaine HCl (50mg). Part A subjects will be asked to perform sensory function assessments, perform motor function assessments and obtain PK samples. Based on the findings of the interim analysis after completion of Part A, the study may stop for futility or proceed to Part B. Part B is a 2-arm study with 120 subjects being randomized 1:1 to either the better performing dosage of EXPAREL from Part A (266mg or 133mg) or 0.25% bupivacaine HCl (50mg).

All eligible subjects will receive Celecoxib 200 mg, orally (PO) pre-operatively within four hours prior to surgery.

Part A: On Day 1, Subjects will be randomized (1:1:1) to receive a sciatic (in the popliteal fossa) nerve block with a single dose of either: EXPAREL 266 mg, EXPAREL 133 mg, or 0.25% bupivacaine HCl (50 mg).

Part B: will continue enrolling with one of the EXPAREL arms (EXPAREL 266 mg arm or EXPAREL 133 mg arm) and the bupivacaine HCl arm. Therefore, the EXPAREL study arm that fails to show efficacy (conditional power less than 30% in the Part A analysis) will be dropped and the study will continue with two study arms. The final analysis will include subjects from both Part A and Part B.

1. If the conditional power of one EXPAREL arm is less than 30% and the other EXPAREL arm is greater than or equal to 30%:

   * The EXPAREL arm with conditional power less than 30% will be dropped in Part B.
2. If both EXPAREL arms have a conditional power greater than or equal to 30%:

   * If the conditional power of the 266 mg EXPAREL arm is more than 10% greater than the conditional power of the 133 mg EXPAREL arm, then the 266 mg EXPAREL arm will be kept and the 133 mg EXPAREL arm will be dropped. Otherwise, the 133 mg EXPAREL arm will be kept and the 266 mg EXPAREL arm will be dropped in Part B.
3. If the conditional power of both treatment arms is less than 30%:

   * The study will stop for futility

All subjects will receive a dose of 1000 mg of intravenous (IV) acetaminophen at the time of surgical incision. All subjects will receive one post-operative dose of 1000 mg IV acetaminophen, administered approximately 8 hours after the first dose (approximately 8 hours after incision). The maximum total dose will not exceed 2000 mg. No additional acetaminophen is permitted after the second IV acetaminophen dose.

Medications will be administered on an as needed (PRN) basis; opioids should not be given on a predetermined schedule.

After 96 hours, the analgesic regimen may be adjusted for each subject individually as deemed appropriate by the physician responsible for postsurgical care.

NRS Pain intensity scores (for pain experiencing in operative foot right now, for the worst pain experienced in the operative foot in the last 24 hours, and for the average pain in the operative foot in the last 24 hours) will be asked from the end of surgery to 96 hours post-surgery at designated timepoints.

Subjects in Part A and Part B will be discharged after the completion of the 168h and 96h assessments, respectively.

For the assessment of adverse events (AEs), SAEs, and concomitant medication use, a follow-up phone call will be made on Post Surgery Day (POD) 14 (±3 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ages 18 or older at screening
2. American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
3. Able to provide informed consent, adhere to the study schedule, and complete all study assessments
4. Primary surgical indication is related to a bunion deformity (i.e., hallux valgus) and subject is scheduled to undergo a distal metaphyseal osteotomy procedure (e.g., Austin procedure as opposed to Lapiplasty, Lapidus bunionectomies or base wedge bunionectomies)
5. Indicated to undergo elective (i.e., not emergency) bunionectomy
6. Body Mass Index (BMI) ≥18 and <40 kg/m2

Exclusion Criteria:

1. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCl, NSAIDs)
2. Concurrent painful physical condition (e.g. arthritis, fibromyalgia, cancer) that may require analgesic treatment with NSAIDs or opioids in the post dosing period for pain that is not strictly related to the foot surgery and which, in the Investigator's opinion, may confound the post dosing assessments
3. Inadequate sensory function of the foot/ankle as assessed by the Investigator
4. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
5. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study
6. Previous participation in an EXPAREL study
7. Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance
8. Currently pregnant, nursing, or planning to become pregnant during the study
9. Clinically significant medical disease that, in the opinion of the Investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction or other conditions that would constitute a contraindication to participation in the study
10. Currently on a neuromodulating agent (e.g., gabapentin, pregabalin [Lyrica], duloxetine [Cymbalta], etc.)
11. Current use of systemic glucocorticoids within 30 days of randomization in this study
12. Use of dexmedetomidine HCl (Precedex®) or clonidine within 3 days of study drug administration
13. Any use of marijuana (including tetrahydrocannabinol (THC) and cannabidiol (CBD)) within 30 days prior to randomization, or planned use during the course of the study
14. Chronic opioid use within 30 days prior to randomization (average ≥30 oral morphine equivalents/day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Nevins, Study Director — Pacira Pharmaceuticals, Inc
Locations (7):
- United States (7):
  - Arkansas Surgical Hospital, North Little Rock, Arkansas
  - Lotus Clinical Research, Pasadena, California
  - Midwest Clinical Research Center, Dayton, Ohio
  - HD Research- First Surgical Hospital, Bellaire, Texas
  - HD Research-Legent Orthopedic Hospital, Carrollton, Texas
  - Houston Heights Hospital, Houston, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz G, Gadsden JC, Gonzales J, Hutchins J, Song J, Brady O, DiGiorgi M, Winston R. A phase 3 active-controlled trial of liposomal bupivacaine via sciatic nerve block in the popliteal fossa after bunionectomy. J Clin Anesth. 2024 Jun;94:111402. doi: 10.1016/j.jclinane.2024.111402. Epub 2024 Feb 9. PMID 38340677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 6 sites between February 2022 and April 2022 for Part A and between April 2022 and July 2022 for Part B. The first participant was enrolled on February 15, 2022 and the last participant was enrolled on July 18, 2022.
Pre-assignment Details: Of 452 screened participants, 185 met inclusion criteria and were randomized to treatment in Part A (66 participants) or Part B (119 participants). Overall results are presented per treatment arm
Groups:
- EXPAREL 266 mg Arm: subjects randomized to this treatment arm received 20 mL (266 mg) EXPAREL mixed with 10 mL saline
  Bupivacaine liposome injectable suspension 266 mg: Sciatic nerve block in the popliteal fossa with EXPAREL 266 mg
- EXPAREL 133 mg Arm: subjects randomized to this treatment arm received 10 mL (133 mg) EXPAREL mixed with 20 mL saline
  Bupivacaine liposome injectable suspension 133 mg: Sciatic nerve block in the popliteal fossa with EXPAREL 133 mg
- Bupivacaine HCl Arm: Subjects randomized to this treatment arm received 20 mL (50 mg) 0.25% bupivacaine hydrochloric acid (HCl) mixed with 10 mL saline
  Bupivacaine HCl: Sciatic nerve block in the popliteal fossa with Bupivacaine HCl
Period: Part A (14 Days)
Arm/Group | EXPAREL 266 mg Arm | EXPAREL 133 mg Arm | Bupivacaine HCl Arm
Started | 22 | 22 | 22
Completed | 21 | 21 | 19
Not Completed | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Failure to meet continuation criteria | 0 | 0 | 1
Period: Part B (14 Days)
Arm/Group | EXPAREL 266 mg Arm | EXPAREL 133 mg Arm | Bupivacaine HCl Arm
Started (Following completion of Part A, an interim analysis was performed before enrollment in Part B was initiated. The dose of EXPAREL evaluated in Part B (133 mg) was determined based on the interim analysis and the 226 mg arm was dropped. The final analysis includes subjects from both Part A and Part B.) | 0 | 59 | 60
Completed | 0 | 59 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of all participants for whom baseline characteristics were measured
Groups:
- Part A: EXPAREL 266 mg Arm: subjects randomized to this treatment arm received 20 mL (266 mg) EXPAREL mixed with 10 mL saline
  Bupivacaine liposome injectable suspension 266 mg: Sciatic nerve block in the popliteal fossa with EXPAREL 266 mg
- Part A + B: EXPAREL 133 mg Arm: subjects randomized to this treatment arm received 10 mL (133 mg) EXPAREL mixed with 20 mL saline
  Bupivacaine liposome injectable suspension 133 mg: Sciatic nerve block in the popliteal fossa with EXPAREL 133 mg
- Part A + B: Bupivacaine HCl Arm: Subjects randomized to this treatment arm received 20 mL (50 mg) 0.25% bupivacaine HCl mixed with 10 mL saline
  Bupivacaine HCl: Sciatic nerve block in the popliteal fossa with Bupivacaine HCl
- Total: Total of all reporting groups
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm | Total
Number analyzed (Participants) | 22 | 81 | 82 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.36 (10.896) | 50.15 (12.823) | 47.24 (11.950) | 48.65 (12.239)
Age, Customized [Count of Participants; unit: Participants]
  <45 Years | 6 | 28 | 30 | 64
  Between 45 and 65 years | 16 | 45 | 47 | 108
  >=65 years | 0 | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 74 | 68 | 163
  Male | 1 | 7 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 26 | 32 | 68
  Not Hispanic or Latino | 12 | 55 | 50 | 117
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 47 | 49 | 112
  Black/African American | 4 | 25 | 28 | 57
  Other | 2 | 9 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 22 | 81 | 82 | 185
ASA classification [Count of Participants; unit: Participants] — The American Society of Anesthesiologists (ASA) physical classification system is a grading system to determine the health of a person before a surgical procedure that requires anesthesia. The ASA classification was performed at baseline.
  Participants
    ASA 1 | 14 | 39 | 54 | 107
    ASA 2 | 8 | 42 | 28 | 78
Body Mass Index [Count of Participants; unit: Participants]
  <25 kg/m^2 | 8 | 21 | 24 | 53
  25 to <30 kg/m^2 | 10 | 27 | 32 | 69
  ≥30 kg/m^2 | 4 | 33 | 26 | 63
Worst pain intensity (NRS) [Mean (Standard Deviation); unit: units on a scale] — Worst pain intensity scores on a numeric rating scale ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, in the last 30 days of baseline. Mean score is provided. The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worse outcome. Population: One participant in the Bupivacaine HCl arm (Part A) discontinued from the study due to an adverse event on Day 1.
  units on a scale
    number analyzed (Participants) | 22 | 81 | 81 | 184
    (all) | 5.4 (3.00) | 5.2 (2.71) | 5.7 (2.59) | 5.5 (2.69)
Average pain intensity (NRS) [Mean (Standard Deviation); unit: units on a scale] — Average pain intensity scores on a numeric rating scale ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, in the last 30 days of baseline. Mean score is provided. The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worse outcome. Population: One participant in the Bupivacaine HCl arm (Part A) discontinued from the study due to an adverse event on Day 1.
  units on a scale
    number analyzed (Participants) | 22 | 81 | 81 | 184
    (all) | 3.9 (2.23) | 3.4 (2.10) | 3.8 (2.33) | 3.7 (2.22)

OUTCOME MEASURES:

1. Primary Outcome: NRS Pain Scores Through 96 Hours Post-surgery
Description: The numeric rating scale pain intensity scores ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, from 0 to 96 hours post-surgery. For each subject, the area under the curve was derived using the trapezoidal rule on the pain scores adjusted for opioid pain medication using the observed and imputed values. Area under the curve started with the first pain assessment obtained after surgery and use all subsequent pain assessments up to 96 hours post-surgery. Pain scores were taken at 5 interval point 0 hours, 24 hours, 48 hours, 72 hours, and 96 hours. There were also unscheduled pain scores measured before opioid consumption also included in the area under the curve calculation. The area under the curve ranged from 0 to 960. Higher scores represent a worse outcome.
Time Frame: 0- 96 hours post-surgery
Population: The analysis was performed on the efficacy analysis set which included all participants in the safety analysis set who underwent the planned surgery and had at least one post-drug administration NRS pain assessment.
Measure: Mean (Standard Deviation); unit: units on a scale*hours
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
Number analyzed (Participants) | 22 | 81 | 82
units on a scale*hours | 342.3 (265.35) | 201.3 (180.05) | 377.4 (188.60)
Statistical Analysis 1: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; The superiority of EXPAREL to bupivacaine hydrochloric acid (HCI) was evaluated using the Efficacy Analysis Set; Test type: Superiority — A one-sided hypothesis test was performed at alpha=0.025 level of significance comparing EXPAREL and bupivacaine HCI; p < 0.00001, ANCOVA; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Mean Difference (Final Values) = -164.0, 95% CI 2-sided [-218.3 to -109.6], Standard Error of Mean 27.74

2. Secondary Outcome: Postsurgical Opioid Consumption Through 96 Hours Post-surgery
Description: Total postsurgical opioid consumption in oral morphine equivalents (OMED) from 0 to 96 hours post-surgery
Time Frame: 0 to 96 hours post-surgery
Population: The analysis was performed on the efficacy analysis set which included all participants in the safety analysis set who underwent the planned surgery and had at least one post-drug administration NRS pain assessment. Results presented for each treatment arm
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams oral morphine equivalents
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
Number analyzed (Participants) | 22 | 81 | 82
milligrams oral morphine equivalents | 32.68 (96.768) | 15.41 (126.781) | 41.62 (83.925)
Statistical Analysis 1: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; The superiority of EXPAREL to bupivacaine hydrochloric acid (HCI) was evaluated using the Efficacy Analysis Set; Test type: Superiority — A one-sided hypothesis test was performed at alpha=0.025 level of significance comparing EXPAREL and bupivacaine HCI; p < 0.00001, ANCOVA; Least square mean difference = 0.39, 95% CI 2-sided [0.28 to 0.55]

3. Secondary Outcome: Opioid-free Subjects Through 96 Hours Post-surgery
Description: Percentage of opioid-free subjects through 96 hours
Time Frame: 0 to 96 hours post-surgery
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
Number analyzed (Participants) | 22 | 81 | 82
percentage of participants | 4.5 | 33.3 | 9.8
Statistical Analysis 1: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p = 0.0003, ANCOVA; Odds Ratio (OR) = 5.04, 95% CI 2-sided [2.01 to 12.62]

4. Secondary Outcome: First Opioid Consumption Post-surgery
Description: Time to first opioid consumption post-surgery
Time Frame: 0 to 96 hours post-surgery
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
Number analyzed (Participants) | 22 | 81 | 82
hours | 16.06 [12.32 to 20.57] | 20.27 [17.13 to 29.98] | 20.68 [19.28 to 24.40]
Statistical Analysis 1: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p = 0.0089, Cox proportional hazards model; Cox proportional hazards model with treatment as main effect and site as categorical and age as continuous covariates; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.45 to 0.93]

5. Secondary Outcome: NRS Pain Scores Post-surgery
Description: Worst and average NRS pain intensity scores at 24h, 48h, 72h, and 96h from the end of surgery
  Worst and average pain intensity scores on a numeric rating scale ranging from 0 to 10, where 0 equals no pain and 10 equals the worst possible pain, from 0 to 24 hours, 24 to 48 hours, 48 to 72 hours, and 72 to 96 hours. Mean scores at each timepoint are provided. The total range is 0 (no pain) to 10 (worst possible pain). Higher values on the scale represent worse outcome.
Time Frame: 0-24 hours, 24-48 hours, 48-72 hours, and 72-96 hours post-surgery
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant discontinuation from the study in Part A.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
Number analyzed (Participants) | 22 | 81 | 82
units on a scale
  Worst pain at 24 hours: number analyzed (Participants) | 22 | 81 | 81
  Worst pain at 24 hours | 6.0 (3.18) | 4.4 (3.13) | 5.3 (3.06)
  Worst pain at 48 hours: number analyzed (Participants) | 21 | 81 | 80
  Worst pain at 48 hours | 6.1 (2.49) | 4.4 (3.14) | 7.3 (2.22)
  Worst pain at 72 hours: number analyzed (Participants) | 21 | 81 | 80
  Worst pain at 72 hours | 4.3 (3.55) | 2.7 (2.87) | 6.1 (2.69)
  Worst pain at 96 hours: number analyzed (Participants) | 21 | 81 | 80
  Worst pain at 96 hours | 4.4 (3.68) | 2.8 (2.84) | 5.1 (2.81)
  Average pain at 24 hours: number analyzed (Participants) | 22 | 81 | 81
  Average pain at 24 hours | 4.7 (2.60) | 2.8 (2.32) | 3.0 (2.58)
  Average pain at 48 hours: number analyzed (Participants) | 21 | 81 | 80
  Average pain at 48 hours | 3.9 (2.74) | 2.9 (2.33) | 4.8 (2.01)
  Average pain at 72 hours: number analyzed (Participants) | 21 | 81 | 80
  Average pain at 72 hours | 3.5 (3.19) | 1.8 (2.05) | 4.1 (2.19)
  Average pain at 96 hours: number analyzed (Participants) | 21 | 81 | 80
  Average pain at 96 hours | 3.2 (3.14) | 1.7 (2.03) | 3.3 (2.10)
Statistical Analysis 1: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p = 0.0296, ANCOVA — Worst pain 0-24 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariate of age; Least square mean difference = -0.8, 95% CI 2-sided [-1.7 to 0.0], Standard Error of Mean 0.44
Statistical Analysis 2: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Worst pain 24-48 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -2.9, 95% CI 2-sided [-3.6 to -2.1], Standard Error of Mean 0.40
Statistical Analysis 3: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Worst pain 48-72 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -3.3, 95% CI 2-sided [-4.1 to -2.5], Standard Error of Mean 0.41
Statistical Analysis 4: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Worst pain 72-96 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -2.1, 95% CI 2-sided [-3.0 to -1.3], Standard Error of Mean 0.43
Statistical Analysis 5: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p = 0.3419, ANCOVA — Average pain 0-24 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -0.1, 95% CI 2-sided [-0.9 to 0.6], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Average pain 24-48 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -1.9, 95% CI 2-sided [-2.5 to -1.3], Standard Error of Mean 0.31
Statistical Analysis 7: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Average pain 48-72 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -2.2, 95% CI 2-sided [-2.8 to -1.6], Standard Error of Mean 0.31
Statistical Analysis 8: Comparison: Part A + B: EXPAREL 133 mg Arm vs Part A + B: Bupivacaine HCl Arm; Test type: Superiority; p < 0.00001, ANCOVA — Average pain 72-96 hours; Main effect of treatment, categorical covariate of pooled Investigator site, and continuous covariates of age; Least square mean difference = -1.5, 95% CI 2-sided [-2.1 to -0.9], Standard Error of Mean 0.31

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the date and time on or after the start date and time of study drug administration through post-operative Day 14
Description: Participants were expected to volunteer information about adverse events that they experienced. In addition, the investigator or designee questioned the patient at each scheduled time point/visit about adverse events and recorded these as well as other adverse events at the time point/visit. Participants experiencing the same adverse events more than once were counted only once at each summary level.
Arm/Group | Part A: EXPAREL 266 mg Arm | Part A + B: EXPAREL 133 mg Arm | Part A + B: Bupivacaine HCl Arm
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/81 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/81 | 1/82
Other Adverse Events (participants affected / at risk) | 13/22 | 42/81 | 45/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: EXPAREL 266 mg Arm (N=22) | Part A + B: EXPAREL 133 mg Arm (N=81) | Part A + B: Bupivacaine HCl Arm (N=82)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: EXPAREL 266 mg Arm (N=22) | Part A + B: EXPAREL 133 mg Arm (N=81) | Part A + B: Bupivacaine HCl Arm (N=82)
Nausea (Gastrointestinal disorders) | 9 (11) | 13 (14) | 19 (19)
Constipation (Gastrointestinal disorders) | 3 (3) | 10 (10) | 16 (16)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (6) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 8 (10) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions include:

* PIs or any other party are not allowed to publish any publication for a period of twelve months following completion of the clinical study report for the trial.
* PIs or any other party shall submit a proposal to the Sponsor for approval to obtain trial results that have not been previously made public and any publication, abstract or paper or other written materials to the trial shall be submitted to the Sponsor at least 60 days prior to submission.

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT05157841/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT05157841/SAP_001.pdf